CLINICAL TRIAL: NCT01548157
Title: A Randomized, Open Label, Single Dose, 2X2 Cross-over Study to Compare Pharmacokinetics Between Rosuvastatin 10mg and Omega-3 1g Co-administration and HCP1007 in Healthy Male Volunteers
Brief Title: Clinical Trial to Evaluate the Effect on the Pharmacokinetic Characteristics of HCP1007 Capsule
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-ROMA-101
Record Dates: First submitted 2012-02-27; First posted 2012-03-08 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: HCP1007; Rosuvastatin; Omega-3
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HCP1007 (Experimental): HCP1007
  Interventions: Drug: HCP1007 / omarco and crestor
- omarco and crestor (Active Comparator): Rosuvastatin plus Omega-3
  Interventions: Drug: HCP1007 / omarco and crestor

INTERVENTIONS:
Drug: HCP1007 / omarco and crestor — HCP1007 / Rosuvastatin plus Omega-3

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics and safety after oral administration of HCP1007 capsules and Rosuvastatin plus Omega-3.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate pharmacokinetics and safety after oral administration of HCP1007 capsules and Rosuvastatin plus Omega-3.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age between 20 and 45
* Informed of the investigational nature of this study and voluntarily agree to participate in this study
* BMI of >20kg/m2 and <26kg/m2 subject

Exclusion Criteria:

* Use of any prescription medication within 14 days prior to Day 1
* Use of any medication within 7 days prior to Day 1
* Participation in another clinical study within 60 days prior to start of study drug administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2012-03; Primary Completion 2012-03 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Area Under Curve(AUC) last | 0,0.5,1,1.5,2,2.5,3,4,5,6,9,12,24,48hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: kyun seop Bae, MD, Ph.D, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea